CLINICAL TRIAL: NCT04098523
Title: Prevalence of Carotid Artery Stenosis and Abdominal Aortic Aneurysms in Brussels: a Population-based Screening Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erik Debing (Other)
Responsible Party: Sponsor-Investigator, Erik Debing, Head of the Department of Vascular Surgery Professor Doctor Erik Debing, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GALSKELA01
Record Dates: First submitted 2019-09-04; First posted 2019-09-23 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Carotid Artery Stenosis; Abdominal Aortic Aneurysm; Epidemiology
Keywords: Carotid Artery Stenosis; Abdominal Aortic Aneurysm; Epidemiology; Stenosis; Population screening
MeSH Terms: conditions — Carotid Stenosis; Aortic Aneurysm, Abdominal; Constriction, Pathologic | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidemiologic screening (Other): All subjects are screened by duplex ultrasound for abdominal aortic aneurysm (AAA) and carotid artery stenosis (CAS). A questionnaire is completed to obtain information on demographic information, risk factors as well as prior treatment for AAA or CAS and current medication. No treatment is given.
  Interventions: Diagnostic Test: Duplex ultrasound

INTERVENTIONS:
Diagnostic Test: Duplex ultrasound — A one-time carotis and abdominal aorta duplex ultrasound will be performed on-site by a skilled site staff to determine the prevalence of, and risk factors associated with, CAS and AAA. A diameter measurement will be performed of the abdominal aorta as well as a determination of the carotid arteries.

SUMMARY:
Both abdominal aortic aneurysm (AAA) and carotid artery stenosis (CAS) are frequent clinical entities, with major morbidity and mortality.

This project obtains robust data on the prevalence of AAA and CAS in the Brussels Capital Region. Using duplex ultrasound, a low invasive examination, we want to obtain information on a vast sample of men and women of the Brussels capital region, starting at the age of 60. With these data we can have a far better view on the Belgian situation of these two main vascular clinical entities. The data can provide insights on if, and how, Belgian public health policy can be improved concerning AAA and CAS.

DETAILED DESCRIPTION:
A population-based screening study to determine the prevalence of carotid artery stenosis (CAS) and abdominal aortic aneurysms (AAA) in the Brussels Capital Region.

The study population is the 60+ inhabitants of the Brussels capital region; recruitment of 4680 subjects. Using duplex ultrasound, a low invasive examination, information is obtained on the abdominal aortic diameter and the degree of stenosis of the carotid bifurcation.

The objective is to determine not only the prevalence of, but also the risk factors associated with CAS and AAA among 60+ Brussels inhabitants. To collect these data, a questionnaire is made including demographic features, associated risk factors, but also previous treatment for AAA or CAS and the current medication of the subject.

Examination is done by one-time duplex ultrasound to perform a diameter measurement of the abdominal aorta and determine the degree of stenosis of the carotid arteries.

Data collection will be done in an electronic case report form, and statistical analysis will be done by a multi-variable logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate is at least 60 years old.
2. Candidate lives in Brussels capital region at the time of study participation.
3. Candidate must sign and date the informed consent form prior to study participation.

Exclusion Criteria:

1. Candidate is suspected of being unable to comply with the study protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3286 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of CAS and AAA among 60+ Brussels inhabitants. | Screening period of 2 years
  Determine the prevalence using echo duplex screening.
Risk factors associated with CAS and AAA among 60+ Brussels inhabitants. | Screening period of 2 years
  Determine the risk factors via a questionnaire:
  * Smoking (ex - current - none)
  * Hypertension (medical history - current)
  * Coronary Artery Disease (history of angina pectoris or myocardial infarction)
  * Diabetes Mellitus (history of diet or medically-treated diabetes - type I or II)
  * History of Cerebro Vascular Disease (stroke or TIA)
  * Family (parents/siblings) history (AAA, CVD, …)
  * Hypercholesterolemia
  * Body weight & length (BMI)
  * COPD

CONTACTS AND LOCATIONS:
Overall Officials: Erik Debing, Prof. Dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No